CLINICAL TRIAL: NCT04619732
Title: A Clinical Pilot Study Investigating the Real-time Dynamics of Glucose, Lactate and Creatinine Concentrations in Marginal Donor Kidneys Undergoing Hypothermic Machine Perfusion
Brief Title: Real-time Monitoring of Kidney Grafts on Hypothermic Machine Perfusion
Acronym: REMO-HYMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Accunea Ltd. (Industry)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REMO-HYMAP 2020
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Transplant;Failure,Kidney
Keywords: creatinine; microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Marginal Kidneys (Experimental): Transplant patients receiving kidneys from deceased marginal donors: aged >= 60, or >= 50 with comorbid renal impairment, hypertension, or cerebrovascular disease.
  Following consent, kidneys will be cold perfused with preserving solution for 2-4 hours as per standard of care at the study centre. During this period, the kidneys will be monitored for creatinine, glucose, and lactate concentrations using three microdialysis probes placed into the tissue, the vein, and the ureter. Data will be blinded to clinicians.
  The probes will be removed at the end of the perfusion period and the organs will be transplanted or discarded according to clinical protocol. If transplanted, the study will monitor the patient's recovery for the first 30 days.
  Interventions: Diagnostic Test: Monitoring biochemical concentrations during cold machine perfusion

INTERVENTIONS:
Diagnostic Test: Monitoring biochemical concentrations during cold machine perfusion — Three microdialysis probes will be introduced into the kidney tissues, the vein and ureter in order to measure creatinine, glucose and lactate while the organ is undergoing cold perfusion prior to transplantation.

SUMMARY:
A significant number of deceased donor kidneys donated for transplantation are not used and are thrown away due to lack of ways of checking their condition and function before the operation. This significantly reduces the number of potentially life saving transplants.

The researchers wish to run a small pilot study to see if it is possible to improve the way transplant kidneys are assessed before transplantation by measuring how well they filter the blood, and how good their metabolism is. The researchers believe this new method will help transplant surgeons make better decisions about which kidneys to use.

This pilot study will look at 10 kidneys obtained from older deceased donors. These kidneys are most at risk of being thrown away because of the condition of the donor they came from. At the hospital, these kidneys are usually put onto a machine which pumps cold preservation solution through them for a couple of hours. This time lets the transplant surgeons see how well or poorly the kidney responds to the flowing fluid.

In this study the research team will do exactly the same, but also insert a small probe less than a millimetre in diameter into the kidney and the vein (draining blood pipe) and urine output to monitor a number of chemicals made by the kidney. The researchers believe that the changing levels of these chemicals will give the surgeons much more information than they have now. This probe is removed when the kidney is transplanted.

Combining these levels with news of how well the patients recover after surgery will allow the research team to design a much larger study to get the right level of information to change the way surgeons choose kidneys and help more transplants happen in the future.

ELIGIBILITY:
Inclusion Criteria:

* All organs to be used in the study must be intended for transplantation and not already rejected/discarded.
* All organs must be sourced from deceased donors through NHSBT in the normal course of clinical activity.
* Kidneys must come from marginal or 'imperfect' donors according to current clinical criteria. This typically indicates an age of 60 and over, or 50 and over with one or more premorbid conditions, including renal impairment, cerebrovascular disease, and hypertension.

Exclusion Criteria:

* Organs from living donors are excluded.
* Organs from young healthy donors are excluded.
* Organs will be excluded if on the assessment of the clinical team they are not suitable for hypothermic machine perfusion. This indicates organs that have arrived with visible defects, or fall well outside the team's standard criteria for clinical acceptability (excessive time in transit, excessive warm ischaemia time, excessive cold ischaemia time, very poor pre-morbid donor condition).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative recovery of kidney function | 30 days post-operatively
  Magnitude of change in patient baseline serum creatinine concentration pre- and post-operatively at 30 days (in umol/L)

SECONDARY OUTCOMES:
Reintervention rate | 30 days post-operatively
  Any need to return the patient to theatre or perform additional procedures following the transplant
Primary non-function | 30 days post-operatively
  Number of participants with no change in serum creatinine concentration from baseline despite transplantation
Delayed graft function | 30 days post-operatively
  Number of days with inadequate graft function following surgery (low urine output, static serum creatinine concentration)
Acute rejection | 30 days post-operatively
  Number of patients experiencing immunological rejection of the organ
Post-operative complications | 30 days post-operatively
  Rates of the most common complications including arterial, venous, or parenchymal thrombosis, ureteric leak or stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios Papalois, MD PhD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share non-anonymised patient data with other researchers.